CLINICAL TRIAL: NCT00789971
Title: A Comparison of a Single Orbital Floor Injection of Triamcinolone Versus Conventional Steroid and Antibiotic Drops Used Post Operatively in Uneventful Phacoemulsification Surgery
Brief Title: Triamcinolone Versus Topical Treatment in Post Operative Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sligo General Hospital (Other)
Responsible Party: Catherine Prendiville, Ophthalmolgy Department, Sligo General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Sligogh
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Ocular Inflammation
Keywords: orbital floor triamcinolone; phacoemulsification; post op inflammation; cmo
MeSH Terms: conditions — Chronic recurrent multifocal osteomyelitis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: triamcinolone acetonide — 40 mg of triamcinolone acetonide given inferotemporally perioperatively during phacoemulsification
  Other Names: Kenelog
Drug: Maxitriol — one month of topical G. Dexamethasone 0.1% with Neomycin sulphate 3500IU/g

SUMMARY:
Cataract extraction is one of the most common operative procedures performed throughout the world. Conventionally, patients are discharged with postoperative drops of steroids and antibiotics or a combination of both. These drops are to be administered for 2-6 weeks depending on individual eye unit protocol. Many patients find the postoperative drops arduous and non-compliance can cause prolonged inflammation and discomfort. Patients with cognitive, physical and visual impairments require assistance from family or community nurses to administer drops. A single perioperative injection of Triamcinolone has been shown to be an effective replacement for drops postoperatively in two previous studies 1, 2.

Aims & objectives

The aim of this study is to see if a single orbital floor injection of Triamcinolone is equivalent to conventional steroid and antibiotic drops used post operatively in uneventful phacoemulsification surgery in treating postoperative inflammation.

DETAILED DESCRIPTION:
This is a prospective randomized control trial of 80 patients undergoing routine phacoemulsification cataract extraction. The patients were randomly assigned to receive the triamcinolone injection or post operative topical treatment of G Maxitriol QDS 1/52 tapering over one month. Forty mg of triamcinolone was injected inferior temporally immediately post operatively prior to undraping the patient in theatre in those randomized to this group. The patients were reviewed at week one and at one month.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated cataract surgery, ability to attend follow appointments at one week and one month

Exclusion Criteria:

* included premorbid ocular pathology including previous ocular inflammation and glaucoma, previous ocular surgery, history of CMO, diabetes, concurrent use of systemic anti-inflammatories including inhaled or topical therapy, history of systemic inflammation, inability to attend follow up appointments at one week and one month, complicated cataract surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
ocular inflammation | one week and one month post op

SECONDARY OUTCOMES:
intraocular pressure | one week and one month post op
cystoid macular oedema | one month post op

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mullaney, FRCOphth, Study Director — Sligo General Hospital
Locations (1):
- Sligo General Hospital, Sligo, Sligo, Ireland

REFERENCES:
- [Background] Paganelli F, Cardillo JA, Melo LA Jr, Oliveira AG, Skaf M, Costa RA; Brazilian Ocular Pharmacology and Pharmaceutical Technology Research Group. A single intraoperative sub-Tenon's capsule triamcinolone acetonide injection for the treatment of post-cataract surgery inflammation. Ophthalmology. 2004 Nov;111(11):2102-8. doi: 10.1016/j.ophtha.2004.04.026. PMID 15522378
- [Background] Negi AK, Browning AC, Vernon SA. Single perioperative triamcinolone injection versus standard postoperative steroid drops after uneventful phacoemulsification surgery: Randomized controlled trial. J Cataract Refract Surg. 2006 Mar;32(3):468-74. doi: 10.1016/j.jcrs.2005.12.102. PMID 16631060